CLINICAL TRIAL: NCT05790109
Title: Operator and Patient Acceptance of Radiofrequency Cautery of the Biopsy Track During Percutaneous Liver, Kidney or Spleen Biopsy Procedures.
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: changed study design to retrospective study, since the study intervention is already in routine clinical practice
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Paul Bernard Shyn, Associate Professor of Radiology, Brigham and Women's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2022P001476
Record Dates: First submitted 2023-03-14; First posted 2023-03-29 (Actual); Last update posted 2025-11-03 (Actual); Status verified 2023-07

CONDITIONS: Bleeding Disorder; Spleen Lesion; Liver Diseases; Kidney Diseases
Keywords: Biopsy; Cautery; Bleeding; Liver; Kidney; Spleen; Hemostasis
MeSH Terms: conditions — Hemostatic Disorders; Liver Diseases; Kidney Diseases; Hemorrhage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- RF biopsy track cautery (Experimental): This study is designed as an open-label, single arm study, wherein all study participants will undergo RF track cautery during percutaneous liver, kidney, or spleen biopsy.
  Interventions: Device: RF track cautery during percutaneous organ biopsy

INTERVENTIONS:
Device: RF track cautery during percutaneous organ biopsy — After biopsy samples are obtained, the physician operator will place a radiofrequency bipolar cautery electrode through the biopsy introducer needle into the biopsy track and cauterize the track using a standardized protocol.

SUMMARY:
The goal of this study is to assess the physician and patient experience of radio frequency (RF) track cautery in patients undergoing needle biopsy of the liver, kidney, or spleen who have one or more risk factors for biopsy-related bleeding. RF track cautery involves inserting a bipolar electrode through the same introducer needle used for the biopsy, and heating the tissues along the path of the biopsy needle to prevent bleeding. This study primarily aims to assess the operator and patient experience during the use of track cautery. Secondary aims are to assess the technical success rate and procedure adverse events. Participants who enroll in the study will undergo track cautery as part of their clinically indicated liver, kidney, or spleen biopsy. After the procedure, they will fill out a brief survey asking about their experience during the procedure. Physician operators who perform track cautery as part of the study will also fill out a survey after each procedure asking about their experience using this technique.

DETAILED DESCRIPTION:
Percutaneous biopsies of abdominal organs (liver, kidney, spleen) are commonly performed procedures and, while generally considered safe, have a small risk of post-biopsy hemorrhage. Bleeding risks of percutaneous biopsy are known to be higher for solid abdominal organs including liver, kidney and spleen, than for abdominal biopsies not involving these organs (for example, peritoneal masses or lymph nodes) Some patients also exhibit an increase in bleeding risk due to alterations in coagulation parameters or platelet number and function, which are known to increase rates of post-biopsy hemorrhage. Existing corrective measures for bleeding diathesis such as blood product transfusions are costly and confer additional risks, and do not address the mechanical tissue and vessel injury that sometimes underlies post-biopsy bleeding. Injection of gelatin sponge or other materials into the biopsy track via the introducer needle, while commonly used, can be cumbersome and imprecise, and has not yet clearly demonstrated a benefit in reducing post-biopsy bleeding in human studies.

High-frequency RF cautery, a technique ubiquitous in modern surgical practice, is routinely used for intraoperative hemostasis. This technique is also routinely used during image-guided percutaneous thermal ablation procedures, where the needle track created by the ablation probe is cauterized during probe retraction. An FDA-cleared bipolar RF cautery device that fits through a 17G biopsy introducer needle is now in clinical use, for the purpose of minimizing bleeding during percutaneous image-guided procedures. This study aims to prospectively study the physician and patient experience of using RF track cautery in patients undergoing percutaneous liver, kidney, or spleen biopsy procedures.

Primary aims of the study are:

* Determine how the use of radiofrequency (RF) track cautery during percutaneous solid organ biopsy affects operator experience.
* Determine how the use of radiofrequency (RF) track cautery during percutaneous solid organ biopsy affects patient experience.

Secondary aims of the study are:

* Determine the technical success rate of RF track cautery during percutaneous solid organ biopsy, defined by successful deployment of the cautery electrode through the biopsy introducer needle and application of radiofrequency current to the biopsy track.
* Monitor adverse events, such as bleeding, during and after biopsy procedures in which RF track cautery is used.

ELIGIBILITY:
Inclusion Criteria:

Patients referred to interventional radiology for clinically indicated liver, kidney, or spleen biopsy for diffuse or focal disease, who also have one or more of the following risk factors for bleeding:

* Coagulopathy (INR ≥ 1.5) or thrombocytopenia (platelets < 50) before correction
* Renal disease with glomerular filtration rate (GFR) < 30 ml/min
* Liver cirrhosis
* Anticoagulant or antiplatelet medications where periprocedural withholding poses
* Competing medical risk, or the urgency of the procedure precludes holding the anticoagulant medications for the standard interval (departmental guidelines).
* Any splenic biopsy
* Hypervascular masses in the liver or kidney
* Renal and liver parenchymal biopsies, which are known to carry a higher risk of bleeding.

Exclusion Criteria:

* Uncorrectable coagulopathy (INR remaining ≥ 2.5) or thrombocytopenia (platelets remaining < 25)
* Pregnancy
* Patients who are not competent to provide their own consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-05-23 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Patient experience during use of radiofrequency track cautery during percutaneous organ biopsy | Within 6 hours after procedure
  Patient experience will be assessed via a questionnaire completed while in the recovery area following their procedure. The patient questionnaire will include questions regarding patient recollection of discomfort related to RF cautery, and whether or not they would be willing to have RF cautery performed again during a future biopsy session, if indicated.
Operator experience during use of radiofrequency track cautery during percutaneous organ biopsy | Within 7 days after procedure
  Operator experience will be assessed via a post-procedure questionnaire (included below) administered to all study operators immediately after they perform each biopsy procedure with RF cautery. The operator questionnaire will consist of a series of questions related to the use of RF cautery, focusing on factors such as ease of use, added procedure time, perceived benefits/detriments, and the operator's perception of associated patient discomfort.

SECONDARY OUTCOMES:
Technical success rate of radiofrequency track cautery during percutaneous organ biopsy | Within 7 days after procedure
  Technical success will be defined by successful deployment of the cautery electrode through the introducer needle into the region sampled by the biopsy needle and application of radiofrequency current for the requisite duration. This will be assessed based on a combination of self-reported technical success by the operator as well as retrospective review of the intraprocedural images by the study investigators.
Adverse events of radiofrequency track cautery during percutaneous organ biopsy | Within 30 days after procedure
  Adverse events will be assessed by recording any major and minor adverse events (including bleeding) that occur during or after biopsy procedures where RF cautery was used.

CONTACTS AND LOCATIONS:
Overall Officials: Paul B Shyn, M.D., Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Minami Y, Hayaishi S, Kudo M. Radiofrequency ablation for hepatic malignancies: is needle tract cauterization necessary for preventing iatrogenic bleeding? Dig Dis. 2013;31(5-6):480-4. doi: 10.1159/000355254. Epub 2013 Nov 21. PMID 24281024
- [Background] Laeseke PF, Winter TC 3rd, Davis CL, Stevens KR, Johnson CD, Fronczak FJ, Webster JG, Lee FT Jr. Postbiopsy bleeding in a porcine model: reduction with radio-frequency ablation--preliminary results. Radiology. 2003 May;227(2):493-9. doi: 10.1148/radiol.2272020173. Epub 2003 Apr 3. PMID 12676970
- [Background] Pritchard WF, Wray-Cahen D, Karanian JW, Hilbert S, Wood BJ. Radiofrequency cauterization with biopsy introducer needle. J Vasc Interv Radiol. 2004 Feb;15(2 Pt 1):183-7. doi: 10.1097/01.rvi.000019398.74740.69. PMID 14963187
- [Background] Lim S, Rhim H, Lee MW, Song KD, Kang TW, Kim YS, Lim HK. New Radiofrequency Device to Reduce Bleeding after Core Needle Biopsy: Experimental Study in a Porcine Liver Model. Korean J Radiol. 2017 Jan-Feb;18(1):173-179. doi: 10.3348/kjr.2017.18.1.173. Epub 2017 Jan 5. PMID 28096727
- [Background] Choi SH, Lee JM, Lee KH, Kim SH, Lee JY, Han JK, Choi BI. Postbiopsy splenic bleeding in a dog model: comparison of cauterization, embolization, and plugging of the needle tract. AJR Am J Roentgenol. 2005 Oct;185(4):878-84. doi: 10.2214/AJR.04.1395. PMID 16177404
- [Background] Song KD, Rhim H, Lee MW, Kang TW, Lim S. A radiofrequency device for tract ablation after liver biopsy: a single-institution human feasibility study. Br J Radiol. 2018 May;91(1085):20170585. doi: 10.1259/bjr.20170585. Epub 2018 Mar 8. PMID 29356562